CLINICAL TRIAL: NCT04064229
Title: ivWatch Sensor: Device Validation for Infiltrated Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ivWatch, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IVW-CLR-CS27-400
Record Dates: First submitted 2019-08-20; First posted 2019-08-21 (Actual); Results first posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-05

CONDITIONS: Infiltration of Peripheral IV Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Infiltrated Tissue (Experimental): The ivWatch Model 400 sensors monitored an IV site during the infiltration of 10 mL of isotonic saline solution. IV sites were placed in the forearm and the dorsal aspect of the hand. The rate of the infiltration ranged between 5 mL/hr to 150 mL/hr.
  Interventions: Device: ivWatch Model 400 with SmartTouch Sensor; Device: ivWatch Model 400 with Fiber Optic Sensor

INTERVENTIONS:
Device: ivWatch Model 400 with SmartTouch Sensor — The ivWatch Model 400 with SmartTouch Sensor monitored the site during the course of the infiltration and issued red and/or yellow notifications if an infiltration was detected.
Device: ivWatch Model 400 with Fiber Optic Sensor — The ivWatch Model 400 with Fiber Optic Sensor monitored the site during the course of the infiltration and issued red and/or yellow notifications if an infiltration was detected.

SUMMARY:
A single arm trial consisting of 98 adult volunteers to assess the safety and efficacy of ivWatch sensors when observing infiltrated tissues at common sites for peripheral IV therapy.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Pass health screen by clinician
* 18 years or older

Exclusion Criteria:

* Fail health screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ivWatch, LLC, Williamsburg, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: IV site
Groups:
- Infiltrated Tissue: The ivWatch Model 400 sensors monitored an IV site during the infiltration of 10 mL of isotonic saline solution. IV sites were placed in the forearm and the dorsal aspect of the hand. The rate of the infiltration ranged between 5 mL/hr to 150 mL/hr.
  ivWatch Model 400: The ivWatch Model 400 monitored the site during the course of the infiltration and issued red and/or yellow notifications if an infiltration was detected.
Period: Overall Study
Arm/Group | Infiltrated Tissue
Started | 99; 198 IV site
Completed | 99; 198 IV site
Not Completed | 0; 0 IV site

BASELINE CHARACTERISTICS:
Population: One case study (participant) was rejected and removed from analysis because there was a protocol error where the IV tubing was not properly connected, and the saline was leaked from the tubing rather than injected at the skin site.
Units Other Than Participants: IV Site
Arm/Group | Infiltrated Tissue
Number analyzed (Participants) | 98
Number analyzed (IV Site) | 196
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 92
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Skin Pigmentation [Mean (Standard Deviation); unit: units on a scale] — Skin pigmentation was scored from 1 to 3 where 1 represents light skin pigmentation, 2 represents medium skin pigmentation, and 3 represents dark skin pigmentation.
  units on a scale | 1.76 (0.84)
Body Mass Index (BMI) [Count of Participants; unit: Participants] — BMI = 703 * weight (lb.) / (height (in.)^2)
  Participants
    Normal (BMI 18.5 to < 25) | 22
    Overweight (BMI 25 to < 30) | 29
    Obese (BMI >= 30) | 47

OUTCOME MEASURES:

1. Primary Outcome: Red Notification Sensitivity to Infiltrated Tissues
Description: The ratio of the number of infiltrated IV sites where the ivWatch Model 400 device issued a red notification to the total number of infiltrated IV sites in the study. All infiltrations were limited to 10 mL of isotonic saline solution.
Time Frame: After each participant has been infiltrated, an expected average of 1 hour
Measure: Mean (95% Confidence Interval); unit: percentage of infiltrations detected
Units Other Than Participants: IV Site
Groups:
- SmartTouch Sensor: ivWatch Model 400 with SmartTouch sensor used to monitor IV site
- Fiber Optic Sensor: ivWatch Model 400 with Fiber Optic sensor used to monitor IV site
Arm/Group | SmartTouch Sensor | Fiber Optic Sensor
Number analyzed (Participants) | 98 | 98
Number analyzed (IV Site) | 98 | 98
percentage of infiltrations detected | 99.0 [94.5 to 100.0] | 99.0 [94.5 to 100.0]

2. Secondary Outcome: Yellow Notification Sensitivity to Infiltrated Tissues
Description: The ratio of the number of infiltrated IV sites where the ivWatch Model 400 device issued a yellow notification to the total number of infiltrated IV sites in the study. All infiltrations were limited to 10 mL of isotonic saline solution.
Time Frame: After each participant has been infiltrated, an expected average of 1 hour
Measure: Mean (95% Confidence Interval); unit: percentage of infiltrations detected
Units Other Than Participants: IV SIte
Arm/Group | SmartTouch Sensor | Fiber Optic Sensor
Number analyzed (Participants) | 98 | 98
Number analyzed (IV SIte) | 98 | 98
percentage of infiltrations detected | 99.0 [94.5 to 100.0] | 99.0 [94.5 to 100.0]

3. Secondary Outcome: Infiltrated Volume When Red Notification Issued
Description: The amount of infiltrated isotonic saline solution when the red notification was issued by the ivWatch Model 400 device.
Time Frame: After each participant has been infiltrated, an expected average of 1 hour
Measure: Median (Standard Deviation); unit: mL
Units Other Than Participants: IV Site
Arm/Group | SmartTouch Sensor | Fiber Optic Sensor
Number analyzed (Participants) | 98 | 98
Number analyzed (IV Site) | 98 | 98
mL | 1.75 (1.45) | 4.33 (2.11)

4. Secondary Outcome: Infiltrated Volume When Yellow Notification Issued
Description: The amount of infiltrated isotonic saline solution when the yellow notification was issued by the ivWatch Model 400 device.
Time Frame: After each participant has been infiltrated, an expected average of 1 hour
Measure: Median (Standard Deviation); unit: mL
Units Other Than Participants: IV Site
Arm/Group | SmartTouch Sensor | Fiber Optic Sensor
Number analyzed (Participants) | 98 | 98
Number analyzed (IV Site) | 98 | 98
mL | 1.66 (1.39) | 3.90 (1.89)

5. Secondary Outcome: Significant Skin Irritation or Disruption to Skin Integrity
Description: The number of IV sites that indicated significant skin irritation or disruption to skin integrity assessed at the end of the study.
Time Frame: After each participant has been infiltrated, an expected average of 1 hour
Measure: Count of Units; unit: IV Site
Units Other Than Participants: IV Site
Arm/Group | SmartTouch Sensor | Fiber Optic Sensor
Number analyzed (Participants) | 98 | 98
Number analyzed (IV Site) | 98 | 98
IV Site | 0 | 0

ADVERSE EVENTS:
Time Frame: A visual assessment of the skin was performed after completing each study. In addition, photos of the skin were captured before and after the study. The time frame of assessment was an expected average of 1 hour after each participant has been infiltrated.
Description: Serious and other (non-serious) adverse events were assessed by the clinician performing the study.
Arm/Group | SmartTouch Sensor | Fiber Optic Sensor
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/99
Other Adverse Events (participants affected / at risk) | 0/99 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT04064229/Prot_SAP_000.pdf